CLINICAL TRIAL: NCT04437485
Title: eIMPACT-DM Pilot Trial: Depression Treatment to Reduce the Excess Diabetes Risk of People With Depression and Prediabetes
Brief Title: eIMPACT-DM Pilot Trial: Depression Treatment to Reduce Diabetes Risk
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jesse Stewart, Professor of Psychology, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1908716624; R21DK123582 (NIH)
Record Dates: First submitted 2020-06-01; First posted 2020-06-18 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Depression; Major Depressive Disorder; Dysthymic Disorder; Depressive Symptoms; Type 2 Diabetes; PreDiabetes; Insulin Resistance
Keywords: Primary Care; Cognitive-Behavioral Therapy; Computer-Based Psychotherapy; Antidepressant Medications
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Dysthymic Disorder; Diabetes Mellitus, Type 2; Prediabetic State; Insulin Resistance | interventions — Cognitive Behavioral Therapy; Primary Health Care; Bupropion; Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- eIMPACT-DM intervention (Experimental): eIMPACT-DM is a 6-month, modernized, collaborative, stepped care intervention consisting of (1) computerized and telephonic cognitive-behavioral therapy for depression and (2) select antidepressant medications included in an algorithm optimized for diabetes risk reduction. It is a collaborative care intervention in which a multidisciplinary team delivers established depression treatments consistent with patient preference. It uses a stepped, flexible, treat-to-target approach that modernizes the IMPACT intervention by harnessing technology to minimize staff and space requirements. Interventions are Good Days Ahead, Problem Solving Treatment in Primary Care, and select FDA-approved antidepressants. The treatment team consists of a depression clinical specialist, a supervising MD with expertise in primary care and IMPACT, and the patients' primary care providers (PCPs).
  Interventions: Behavioral: Good Days Ahead (GDA); Behavioral: Problem Solving Treatment in Primary Care (PST-PC); Drug: Antidepressant Medications
- Active Control (Active Comparator): Active Control (AC) consists of depression education (study staff), symptom monitoring (study staff), and primary care for depression (clinical staff).
  Interventions: Other: Active Control

INTERVENTIONS:
Behavioral: Good Days Ahead (GDA) — GDA (Empower Interactive) is an empirically supported, HIPAA compliant, computerized CBT for depression appropriate for primary care patients and people with little computer experience. GDA uses an interactive, multimedia format to deliver 9 45-minute sessions, the structure and content of which mirror face-to-face CBT. General topics include identifying and modifying automatic thoughts, using behavioral activation and other behavioral methods, identifying and modifying schemas, using effective coping strategies, and employing other core CBT methods. GDA is empirically supported - it is acceptable to patients, achieves superior depression outcomes to waitlist comparators, and yields equivalent (noninferior) depression outcomes to standard face-to-face CBT. To minimize time/transportation barriers, GDA sessions occur at the PI's lab or a location with internet access selected by the patient (patient's, family member's, or friend's home).
  Other Names: Cognitive-Behavioral Therapy (CBT); Internet Psychotherapy
  Arms: eIMPACT-DM intervention
Behavioral: Problem Solving Treatment in Primary Care (PST-PC) — PST-PC is an established, manualized, empirically supported CBT developed for primary care. During the 6-10 30-minute sessions, patients are taught skills for solving problems contributing to depression. We will deliver PST-PC by phone, which has been found to be feasible and efficacious.
  Other Names: Cognitive-Behavioral Therapy (CBT); Telephonic Psychotherapy
  Arms: eIMPACT-DM intervention
Drug: Antidepressant Medications — We first considered all FDA-approved antidepressants and excluded those with weight gain effects (tricyclics, paroxetine, mirtazapine) and those rarely used in primary care (MAOIs). Then, we used existing evidence to inform the structure. We made bupropion (an aminoketone) and fluoxetine (an SSRI) our first-line and second-line antidepressants, as meta-analyses indicate that their use is associated with weight loss. We made other SSRIs (escitalopram, sertraline) and SNRIs (desvenlafaxine, duloxetine, venlafaxine) our third-line antidepressants, given their negligible effects on weight. Our team will make recommendations to the patient's PCP, who will write prescriptions. Our team and the PCP will then collaboratively manage pharmacotherapy.
  Other Names: Bupropion; Selective Serotonin Reuptake Inhibitors (SSRIs); Serotonin-Norepinephrine Reuptake Inhibitors (SNRIs)
  Arms: eIMPACT-DM intervention
Other: Active Control — (1) The graduate research assistant (RA) will have a 50-minute call with AC patients to review depression materials. The RA will provide a list of Eskenazi Health mental health services and will encourage patients to follow-up with their PCP. We will then send an electronic health record message to the PCP encouraging them to address their patient's depression, note that there are no care restrictions, and provide the same list of services. (2) The RA will call AC patients every 4 weeks to assess depressive symptoms and will notify clinical staff to encourage additional care when indicated. (3) AC patients will receive current primary care for depression. The Eskenazi Health primary care clinics utilize a team care approach, with PCPs supported by embedded behavioral health clinicians and affiliated psychiatrists.
  Arms: Active Control

SUMMARY:
This pilot randomized controlled trial seeks: (1) to determine the preliminary efficacy of our modernized collaborative care intervention for depression in improving the diabetes risk markers of hemoglobin A1c and insulin resistance and (2) to explore whether somatic depressive symptoms - i.e., hyperphagia (increased appetite/weight) and/or hypersomnia (increased sleep) - moderate the effect of the eIMPACT-DM intervention on diabetes risk markers.

DETAILED DESCRIPTION:
Diabetes affects 31 million (12%) U.S. adults, and another 82 million (34%) adults have prediabetes, a precursor to diabetes. The ramifications of diabetes are grave and include cardiovascular disease, disability, and death. While these statistics highlight the importance of diabetes prevention, current approaches have only partial effectiveness. This has created a clear need to identify new primary prevention targets and approaches for diabetes, and depression and depression treatment are strong candidates in this regard. Over 20 years of evidence indicates that depression is an independent, clinically important, robust, biobehaviorally plausible, and modifiable risk factor for diabetes. However, research has yet to determine whether depression treatment can prevent the development of diabetes in people with prediabetes. Given that depression is still receiving limited attention in settings where diabetes prevention occurs (e.g., primary care), there is a large cohort of patients with an underdetected or undertreated diabetes risk factor (depression). This status quo and the strong state of the depression-to-diabetes science create the need for a pilot randomized controlled trial to evaluate the utility of depression treatment as a new diabetes prevention strategy. Thus, we propose a pilot RCT of 64 primary care patients (50% minority) with a depressive disorder and prediabetes. Patients will be randomized to 6 months of eIMPACT-DM (intervention) or Active Control (comparator). eIMPACT-DM is our modernized collaborative stepped care intervention consisting of (1) computerized and telephonic cognitive-behavioral therapy for depression and (2) select antidepressant medications included in an algorithm optimized for diabetes risk reduction. Our preliminary data establish the feasibility and antidepressive efficacy of eIMPACT-DM. The Active Control consists of depression education, symptom monitoring, and primary care for depression. Our primary aim is to determine the preliminary efficacy of eIMPACT-DM in improving the diabetes risk markers of hemoglobin A1c (primary outcome) and insulin resistance (secondary outcome). Our exploratory aim is to explore whether somatic depressive symptoms - i.e., hyperphagia (increased appetite/weight) and/or hypersomnia (increased sleep) - moderate the effect of eIMPACT-DM on diabetes risk markers. A positive pilot trial would pave the way to an R01-level RCT by: (1) generating critical proof-of-concept data (eIMPACT-DM can improve A1c) to support the premise of the definitive trial; (2) providing preliminary effect sizes for eIMPACT-DM on diabetes risk markers to help justify future power analyses; (3) identifying a potentially important moderator of eIMPACT-DM efficacy that may need to be incorporated into the definitive trial. Ultimately, demonstrating that depression treatment reduces diabetes risk would identify a novel target (depression) for diabetes prevention efforts, and it would equip healthcare providers with a new practical, scalable, and disseminable intervention (eIMPACT-DM) to help lower diabetes risk for a large cohort of high-risk patients. These practice changes should translate into reduced diabetes morbidity, mortality, and costs.

ELIGIBILITY:
Inclusion Criteria:

* Current primary care patient in Eskenazi Health
* Age ≥18 years
* Depressive disorder at screening
* Prediabetes at screening

Exclusion Criteria:

* History of type 1 or type 2 diabetes
* Major inflammatory conditions: HIV/AIDS, chronic kidney disease, systemic inflammatory disease (e.g., rheumatoid arthritis, lupus, Crohn's disease, and ulcerative colitis), or active cancer/current cancer treatment
* Current pregnancy
* Severe cognitive impairment
* Acute risk of suicide
* History of bipolar disorder or psychosis or current use of an atypical antipsychotic medication:
* Participation in our prior eIMPACT Trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse C Stewart, PhD, Principal Investigator — Indiana University-Purdue University Indianapolis (IUPUI)
Locations (1):
- IUPUI Department of Psychology, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- eIMPACT-DM Intervention: eIMPACT-DM is a 6-month, modernized, collaborative, stepped care intervention consisting of (1) internet and telephonic CBT for depression and (2) select antidepressant medications in an algorithm optimized for diabetes risk reduction. A multidisciplinary team delivers established depression treatments consistent with patient preference. Good Days Ahead (GDA; MindStreet, Inc.) is an empirically supported internet CBT for depression that uses an interactive, multimedia format to deliver 9 45-minute sessions, the structure and content of which mirror face-to-face CBT. GDA sessions occurred at a location with internet access selected by the patient or the PI's lab. Problem Solving Treatment in Primary Care (PST-PC) is an empirically supported CBT. During the 6-10 30-minute sessions, patients are taught skills for solving problems contributing to depression. We delivered PST-PC by phone. Regarding medications, we first considered all FDA-approved antidepressants and excluded those with weight gain effects and those rarely used in primary care. We then made bupropion and fluoxetine our first-line and second-line antidepressants, given their association with weight loss. We made other SSRIs (escitalopram, sertraline) and SNRIs (desvenlafaxine, duloxetine, venlafaxine) our third-line antidepressants, given their negligible effects on weight. Our team made recommendations to the patient's PCP, who wrote prescriptions. Our team and the PCP collaboratively managed pharmacotherapy.
Period: Overall Study
Arm/Group | eIMPACT-DM Intervention | Active Control
Started | 24 | 22
Completed | 21 | 18
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | eIMPACT-DM Intervention | Active Control | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.7 (11.8) | 50.7 (10.4) | 49.6 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 16 | 36
  Male | 4 | 6 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 17 | 33
  White | 4 | 4 | 8
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 22 | 46
Depressive Symptoms [Mean (Standard Deviation); unit: Score on a scale] — Participants completed the reliable and valid Hopkins Symptom Checklist-20 (SCL-20) to assess depressive symptoms. Total scores (mean of items responses, range: 0-4) were computed, with higher scores indicating greater depressive symptoms.
  Score on a scale | 1.82 (0.83) | 1.73 (0.91) | 1.78 (0.91)
Hemoglobin A1c [Mean (Standard Deviation); unit: % (percentage of total hemoglobin)] — Fasting blood samples were collected, and whole blood and plasma aliquots were frozen. Hemoglobin A1c will be measured by a standard method. A1c is the primary outcome because: (1) it is the gold standard measure of glycemia and a common surrogate endpoint, (2) it strongly predicts future diabetes, (3) interventions decreasing A1c improve clinical diabetes endpoints, and (4) diabetes prevention interventions targeting glycemic control result in lower rates of progression from prediabetes to type 2 diabetes. Higher hemoglobin A1c values indicate greater diabetes risk. Population: Values are from observed dataset. 39 out of 46 participants had observed data.
  % (percentage of total hemoglobin)
    number analyzed (Participants) | 21 | 18 | 39
    (all) | 4.97 (0.44) | 4.91 (0.32) | 4.94 (0.38)
HOMA-IR score [Mean (Standard Deviation); unit: HOMA-IR index] — Higher HOMA-IR scores indicate greater insulin resistance. Homeostatic Model of Assessment-Insulin Resistance (HOMA-IR) scores were derived from fasting glucose and insulin values measured by standard assays. HOMA-IR score is an established index of insulin resistance that correlates highly with the more invasive euglycemic clamp and is appropriate for assessing change. Higher HOMA-IR scores indicate greater insulin resistance. Population: Values are from observed dataset. 39 out of 46 participants had observed data.
  HOMA-IR index
    number analyzed (Participants) | 21 | 18 | 39
    (all) | 2.99 (1.69) | 2.10 (0.97) | 2.58 (1.46)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c at 6 Months
Description: Fasting blood samples were collected, and whole blood and plasma aliquots were frozen. Hemoglobin A1c will be measured by a standard method. A1c is the primary outcome because: (1) it is the gold standard measure of glycemia and a common surrogate endpoint, (2) it strongly predicts future diabetes, (3) interventions decreasing A1c improve clinical diabetes endpoints, and (4) diabetes prevention interventions targeting glycemic control result in lower rates of progression from prediabetes to type 2 diabetes. Higher hemoglobin A1c values indicate greater diabetes risk.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: % (percentage of total hemoglobin)
Arm/Group | eIMPACT-DM Intervention | Active Control
Number analyzed (Participants) | 21 | 18
% (percentage of total hemoglobin) | 4.94 (0.47) | 4.88 (0.38)
Statistical Analysis 1: Comparison: eIMPACT-DM Intervention vs Active Control; Test type: Superiority; p = 0.64, ANCOVA; ANCOVA models were run on post-treatment outcome level adjusting for baseline somatic depressive symptoms group (a stratification variable)

2. Secondary Outcome: Homeostatic Model of Assessment-Insulin Resistance (HOMA-IR) Score at 6 Months
Description: Higher HOMA-IR scores indicate greater insulin resistance. Homeostatic Model of Assessment-Insulin Resistance (HOMA-IR) scores were derived from fasting glucose and insulin values measured by standard assays. HOMA-IR score is an established index of insulin resistance that correlates highly with the more invasive euglycemic clamp and is appropriate for assessing change. Higher HOMA-IR scores indicate greater insulin resistance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: HOMA-IR index
Arm/Group | eIMPACT-DM Intervention | Active Control
Number analyzed (Participants) | 21 | 18
HOMA-IR index | 3.48 (2.16) | 2.38 (0.93)
Statistical Analysis 1: Comparison: eIMPACT-DM Intervention vs Active Control; Test type: Superiority; p = 0.046, ANCOVA; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Depressive Symptoms
Description: Participants completed the reliable and valid Hopkins Symptom Checklist-20 (SCL-20) to assess depressive symptoms. Total scores (mean of items responses, range: 0-4) were computed, with higher scores indicating greater depressive symptoms.
Time Frame: 6 months
Population: Missing data was handled using within subject mean imputation when < 25% of the data was missing.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | eIMPACT-DM Intervention | Active Control
Number analyzed (Participants) | 20 | 18
Score on a scale | 1.11 (0.73) | 1.58 (0.89)
Statistical Analysis 1: Comparison: eIMPACT-DM Intervention vs Active Control; Test type: Superiority; p = 0.09, ANCOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: The adverse event monitoring period for each participant was 6 months, corresponding to the time from each participant's pre-treatment visit (i.e., randomization date) to the completion of their post-treatment visit.
Arm/Group | eIMPACT-DM Intervention | Active Control
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22
Other Adverse Events (participants affected / at risk) | 1/24 | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | eIMPACT-DM Intervention (N=24) | Active Control (N=22)
Blood pressure above the call order levels (Cardiac disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT04437485/Prot_SAP_000.pdf
  • Informed Consent Form (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/85/NCT04437485/ICF_001.pdf